CLINICAL TRIAL: NCT03874338
Title: Studies on the Effects of Colchicine on Neutrophil Biology in Acute Myocardial Infarction: A Substudy of the CLEAR SYNERGY (OASIS 9) Trial
Brief Title: CLEAR SYNERGY Neutrophil Substudy
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Population Health Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-01323; 1R01HL146206 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neutrophils.Hypersegmented | Bld-Ser-Plas; STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colchicine
  Interventions: Drug: Colchicine Pill
- Placebo
  Interventions: Drug: Colchicine Pill

INTERVENTIONS:
Drug: Colchicine Pill — Participants in the main CLEAR SYNERGY trial are randomized to colchicine/spironolactone versus placebo in a 2x2 factorial design. The substudy is interested in the evaluation of biospecimens obtained from patients in the colchicine vs placebo group.

SUMMARY:
CLEAR SYNERGY is an international multi center 2x2 randomized placebo controlled trial of colchicine and spironolactone in patients with STEMI. Subjects enrolled in the main CLEAR SYNERGY trial will be asked to participate in this sub study (n=670) to undergo:

1. Evaluation of markers of neutrophil activity at randomization (baseline) and 3 months follow-up in the colchicine versus placebo groups, and;
2. Examination of clinical and genetic factors that determine heterogeneity of treatment response and distinguish colchicine responders from non- responders.

Participants undergo a blood draw at baseline and 3 months follow-up as part of the main trial, and participants who also participate in this sub study will have an additional 2 tablespoons of blood drawn.

The sub study objectives are to:

1. Assess the effect of colchicine on neutrophil activation in response to STEMI.
2. Examine clinical and genetic factors that determine heterogeneity of treatment response anddistinguish colchicine responders from non- responders.
3. Explore the derivation of a risk score that includes markers of neutrophil activity and is associated with adjudicated MACE over 3 years after STEMI, and assess the impact of colchicine on the relation between this risk score and MACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are randomized to the drug RCT portion of the CLEAR SYNERGY (OASIS 9) trial will be eligible for participation in this Neutrophil biomarker substudy.

Exclusion Criteria:

* Use of anti-inflammatory agents (except aspirin)
* Active infection

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are randomized to the drug RCT portion of the CLEAR SYNERGY (OASIS 9) trial will be eligible for participation in this Neutrophil biomarker substudy. These are patients who present with STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
soluble L-selectin | between baseline and 3 months
  Change in soluble L-selectin between baseline and 3 mo after STEMI in the placebo vs. colchicine groups.

SECONDARY OUTCOMES:
Other soluble markers of neutrophil activity | between baseline and 3 months
  Other markers of neutrophil activity will be evaluated at baseline and 3 months after STEMI (myeloperoxidase, matrix metalloproteinase-9, neutrophil gelatinase-associated lipocalin, neutrophil elastase, intercellular/vascular cellular adhesion molecules)
Markers of systemic inflammation | between baseline and 3 months
  Markers of systemic inflammation will be evaluated at baseline and 3 months after STEMI (high sensitive CRP, IL-1β)
Neutrophil-driven responses that may further propagate injury | between baseline and 3 months
  Neutrophil-driven responses that may further propagate injury will be evaluated at baseline and 3 months after STEMI (neutrophil extracellular traps, neutrophil-derived microparticles)

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No